CLINICAL TRIAL: NCT06960135
Title: Predictors of Trifecta Achievement in Open and Laparoscopic Partial Nephrectomy for Localized Renal Tumors
Brief Title: Trifecta Achievement in Open and Laparoscopic Partial Nephrectomy
Acronym: Trifecta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Omar Ahmad Bakheet, Assistant Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVU-MED-URO016-2-22-5-400
Record Dates: First submitted 2025-04-22; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Trifecta Achievement; Pentafecta Achievement
Keywords: Laparoscopic, Partial Nephrectomy; Trifecta, Pentafecta Achievement; Renal Tumors
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open partial nephrectomy (Active Comparator): open partial nephrectomy
  Interventions: Procedure: open partial nephrectomy
- laparoscopic partial nephrectomy (Active Comparator): laparoscopic partial nephrectomy
  Interventions: Procedure: laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: open partial nephrectomy — open partial nephrectomy
  Arms: open partial nephrectomy
Procedure: laparoscopic partial nephrectomy — laparoscopic partial nephrectomy
  Arms: laparoscopic partial nephrectomy

SUMMARY:
Background: Partial nephrectomy (PN) is a reference standard for the management of the cT1 renal mass, primarily due to better preservation of renal function. The aim of this work was to determine trifecta outcomes of open PN (OPN) and laparoscopic PN (LPN) and identify predictive factors for trifecta achievement to evaluate surgical performance, including negative surgical margins, absence of severe surgical complications, and ischemia time less than 25 minutes.

Objectives: this study pointing to determine trifecta outcomes of OPN and LPN and to identify predictive factors for trifecta achievement to evaluate surgical performance, including negative surgical margins, absence of severe surgical complications, and Ischemia time less than 25 Minutes.

DETAILED DESCRIPTION:
Methods: This prospective, randomized study was carried out on 35 patients with clinical T1 N0M0 renal tumors. Patients were divided into two groups: Group A (n=38): underwent OPN and group B (n=32): underwent LPN.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are fit for surgery.

  * Patients with renal tumor who are indicated for partial nephrectomy

Absolute:

1. Solitary kidney.
2. Bilateral renal tumor.
3. CDK.

Relative:

1. Abnormal contralateral kidney (nephropathy, nephrolithiasis, trauma).
2. Metabolic disease associated with renal failure (DM, hypertension).
3. Genetic syndrome with tumor multifocality (VHL syndrome). Elective

1. Clinical T1N0M0 Tumor. 2. Peripheral tumor.

Exclusion Criteria:

* • Patients who are unfit for surgery and who's unfit for laparoscopy.

  * Patients who are contraindicated for partial nephrectomy. As severe and irreversible coagulopathy. Patients who are indicated for radical nephrectomy (extensive tumor, metastatic tumor).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Predictors of Trifecta Achievement in Open ald Laparoscopic Partial Nephrectomy for Localised Renal Tumors | 2 years
  Trifecta achievement is defined as the combination of (1) negative surgical margins, (2) absence of perioperative complications classified as Clavien-Dindo grade III or higher, and (3) warm ischemia time ≤25 minutes.
  factors affecting trifecta achievement among variables including tumor complexity score, patient comorbidities, BMI, surgical approches, special habbites, age or gender.

SECONDARY OUTCOMES:
Pentafecta Achivement | 2 yrs
  Pentafecta achievement is defined as the combination of:
  1. negative surgical margins,
  2. absence of major perioperative complications (Clavien-Dindo grade ≥III),
  3. warm ischemia time ≤25 minutes,
  4. ≥90% preservation of preoperative estimated glomerular filtration rate (eGFR), and
  5. no progression to a higher CKD stage at 12 months postoperative follow-up. Data will be collected from surgical, pathological, and clinical records. Predictors of Pentafecta achievement will be analyzed using multivariable logistic regression.

CONTACTS AND LOCATIONS:
Locations (1):
- SVU hospital, Qena, Egypt, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided